CLINICAL TRIAL: NCT05879679
Title: Pilot Study on the Validity of the Metacognitive Hub Model of Craving in Bulimia Nervosa (BN) and Binge Eating Disorders (BED)
Acronym: MetaBou
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Université de Nantes (Other); Centre d'expertise Poids, Image et Alimentation (CEPIA) (Unknown); Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Sylvain Iceta, Associate professor, Laval University
Other Study IDs: 2024-4019, 22336
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder
Keywords: craving; addiction; metacognition; neurocognition
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Binge Eating Disorder: Participants with a binge eating disorder (DSM-5 criteria)
  Interventions: Behavioral: Food craving induction
- Bulimia Nervosa: Participants with a bulimia nervosa (DSM-5 criteria)
  Interventions: Behavioral: Food craving induction

INTERVENTIONS:
Behavioral: Food craving induction — Standardized craving induction procedure will be used, based on exposure to food-related images (https://www.lippc2s.fr/food-cal-pictures/). Craving intensity will be measured by visual analogic scale before and after the induction sequence.

SUMMARY:
Craving is defined as an irrepressible urge to consume certain products and represents one of the key factors in severe substance use disorders, as illustrated by its recent inclusion as a diagnostic criterion in the most recent fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM 5). However, the pathophysiological models of craving remain debated.

The "metacognitive hub model", a conceptual, experimental and clinical approach to craving, proposes that craving should be considered as the embedded consequence of the interaction between three components (the reflexive, automatic and interoceptive systems), each of which has an implicit and explicit element. This model links the three components by suggesting that metacognitive abilities, the ability to understand one's own cognitive functioning, may be a skill of individuals that allows them to make the three sub-components explicit or not.

To date, the conception of eating disorders is increasingly similar to that of addictive disorders. Indeed, there is growing evidence that the symptomatology of bulimia nervosa and binge eating disorder can be considered in part as an "food addiction" and would fit the diagnostic criteria of an addictive disorder. Bulimia nervosa is an eating disorder (DSM 5) characterized by a cycle of binge eating and compensatory behaviors such as self-induced vomiting that tend to negate or compensate for the effects of the binge eating. Binge eating disorder (DSM 5) is characterized by a cycle of binge eating, but without the compensatory behaviors seen in bulimia nervosa. In addition, there are common neurological aspects as well as similar cognitions between these eating disorders and addictive disorders. Given the importance of craving in addictive pathology, it seems essential to address this issue in bulimia nervosa and binge eating disorder. The cognitive difficulties of patients with bulimia nervosa and binge eating disorder, which are close to the difficulties observed in patients with addictive behaviors, suggest that the "metacognitive hub model" could provide a clear and measurable theoretical framework of the different dimensions of craving.

The overall objective of this project is to explore the relationship between the level of craving induced by food picture exposure and the level of impairment of the reflexive, automatic, interoceptive, and metacognitive systems in women with bulimia nervosa and binge eating disorder and to compare these impairments according to the nature of the eating disorder (i.e., binge eating versus bulimia nervosa).

Our hypotheses are:

1. the induction of food craving will affect the reflexive, automatic, and interoceptive systems of patients with bulimia nervosa and binge eating disorder.
2. the magnitude of the effect of food craving induction on implicit craving and explicit craving will be modulated by the participants' metacognitive abilities.

ELIGIBILITY:
Inclusion Criteria:

* have been medically diagnosed with binge eating disorder or bulimia nervosa
* fluent in french
* able to consent

Exclusion Criteria:

* co-morbid substance use disorder,
* pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants consulted by specialized psychiatrist at IUCPQ Participants who have already participated in a research project and have agreed to be contacted for other projects Participants recruited via the ANEB and Maison l'Éclaircie mailing lists and via an ad on social networks.
  Participants receiving care at the CEPIA or on the CEPIA waiting list.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Attention Network Test (ANT) | 1 hour (after food craving induction)
  The ANT is a task designed to test three attentional networks in children and adults: alerting, orienting, and executive control
Dot Probe Task | 1 hour (after food craving induction)
  To test and measure selective attention
Water load task | 1 hour (after food craving induction)
  This task was originally developed to induce gastric distension and assess gastrointestinal symptoms in patients with functional digestive disorders. This task stimulates the stomach using a natural distension stimulus (i.e., water ingestion) and without the complex hormonal response of a caloric meal.
Live metacognition | 1 hour (after food craving induction)
  "live" metacognitive assessment will be done by asking the participants to rate their level of confidence on a visual analog scale ranging from 0% (I just guessed) to 100% (completely confident) for each items.
Avoidance/Approach task adapted for food craving | 1 hour (after food craving induction)
  In this task, participants are asked to move a joystick that simulates the movement of the food represented in the image. The joystick movements are accompanied by a zoom effect that increases the illusion of movement.

SECONDARY OUTCOMES:
Beck Depression Inventory II (BDI-II) | Baseline
  Minimum score : 0; Maximun score : 63; Higher scores mean a worse outcome.
State-Trait Anxiety Inventory (STAI) | Baseline
  The questionnaire includes two scales (20 items) consisting of a total of 40 questions. For each scale the minimum score is 0 and the maximun score is 80. Higher scores mean a worse outcome.
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline
  The measure provides four attitudinal subscale scores: Restraint (5 items), Eating Concern (5 items), Shape Concern (8 items), and Weight Concern (5 items). An overall Global score is the mean of the four subscale scores. Responses are on a 7-point ordinal response; minimum score : 0, maximun score: 6; higher scores mean a worse outcome.
Food Craving Questionnaire State (FCQ-S) | Baseline
  Minimum : 15; Maximun : 75; Higher scores mean a worse outcome.
Food Craving Questionnaire Trait (FCQ-T) | Baseline
  Minimum : 39; Maximun : 234; Higher scores mean a worse outcome.
Visual Analogic Scale of craving | Baseline, at 1 hour (after craving induction), at 3 hours (end of the session_
  It represents a continuous visual progression of craving from one extreme to another, from "no craving at all" to "extreme and uncontrollable craving," with patients stating the intensity of their current craving between these two extremes.
Schedule for the Assessment of Insight in Eating Disorders (SAI-ED) | Baseline
  Interview-based scale for the multidimensional assessment of insight in eating disorders. It includes three categories: illness awareness, symptom awareness, and treatment engagement. Minimum score : 0, maximun score: 29; Higher scores mean a better outcome.
Difficulties in Emotional Regulation Scale (DERS- 18) | Baseline
  Minimum score : 18, maximun score : 90; Higher scores mean a worse outcome.
Attentional Control Scale (ACS) | Baseline
  Minimum score : 20, maximun score : 80; Higher scores mean a better outcome.
Body Awareness Questionnaire (BAQ) | Baseline
  Minimum score: 18; Maximun score: 126; Higher scores mean a better outcome.

OTHER OUTCOMES:
Age | Baseline
Gender | Baseline
Biological sex | Baseline
Weight | Baseline
Height | Baseline
Body Mass Index (BMI) | Baseline
  Weight / Height2
Waist and hips circumferences | Baseline
  in cm
Menopausal status or contraception | Baseline
Socio-professional category | Baseline
  Number of participants per socioprofessional category as defined by statistic canada
Medical history and concomitant treatment | Baseline
  Rates of various associated diseases (e.g., cardiovascular, digestive disorders). Type of medications (antidepressants, antipsychotics, hypotensive drugs) and their rates.
Ethnic origin | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Iceta, MD, PhD, Principal Investigator — Fondation IUCPQ; Valentin Flaudias, Psy, PhD, Study Chair — Université de Nantes
Locations (3):
- Canada (2):
  - Centre d'expertise Poids, Image et Alimentation (CEPIA), Québec
  - IUCPQ, Québec
- Université de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided